CLINICAL TRIAL: NCT03463564
Title: Effects of Insulin Pump Versus Multiple Daily Injections of Insulin on Glycemic and Metabolic Control in Type 1 Diabetic Patients Transitioned to the Adult Center: the Management and Technology for Transition Study (METRO)
Brief Title: Insulin Pump vs Multiple Daily Injections of Insulin and Glyco-metabolic Control in Type 1 Diabetic Patients
Acronym: METRO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Katherine Esposito, Full Professor of Endocrinology and Metabolism, Head of Diabetes Unit, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24012014-33
Record Dates: First submitted 2018-02-19; First posted 2018-03-13 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; transition; CSII; MDI; glycemic control; glucose variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems

ARMS (2):
- Insulin pump (Active Comparator): Insulin Pump with rapid acting insulin analog lispro
  Interventions: Device: Insulin pump
- Insulin injections (Active Comparator): Four injections of insulin daily consisting in three bolus of a rapid-acting analog lispro or aspart before breakfast, lunch and dinner and one injection at bed-time of basal insulin glargine or degludec
  Interventions: Drug: Insulin injections

INTERVENTIONS:
Device: Insulin pump — Continuous subcutaneous insulin infusion consisting of the delivery of insulin lispro as basal rate and boluses administered before meals.
  Other Names: CSII
  Arms: Insulin pump
Drug: Insulin injections — Four injections of insulin daily consisting in three bolus of a rapid-acting analog lispro or aspart before breakfast, lunch and dinner and one injection of insulin glargine or degludec at bed-time of basal insulin
  Other Names: MDI
  Arms: Insulin injections

SUMMARY:
The transition from the Pediatric clinic to the adult care is a challenging period for young adults with type 1 diabetes, due to the high risk of poor glycemic control. Achieving the glycemic target without hypoglycemia and/or large glucose excursions is of paramount importance for type 1 diabetic patients, who have high variability of daily glucose levels . Both insulin pump therapy and multiple daily injections of insulin are recommended strategy to achieve glycemic control in type 1 diabetes; however, no studies investigated the effects of insulin pump vs insulin injections on glycol-metabolic outcomes in the transition phase. The aim of this study was to evaluate the effects of continuous subcutaneous insulin infusion (CSII) therapy, as compared with multiple daily injections of insulin (MDI), on glycemic and metabolic control, in young type 1 diabetic patients transitioned to the adult diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* T1DM for at least 12 months
* persistent HbA1c levels ≥ 7.5% (58 mmol/mol) despite optimized education therapy,
* recurrent severe hypoglycemic episodes or high glucose variability
* willingness to wear the insulin pump

Exclusion Criteria:

* previous use of insulin pump
* pregnancy or planning to become pregnant in the next 2 years,
* lack of ability to use the study devices
* history of severe chronic diseases
* recent or concomitant use of corticosteroids
* drug or alcohol abuse
* psychiatric complaints that interfere with the correct use of the devices

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c change | Baseline, 6 months, 12 months, 24 months
  Within and between groups difference in HbA1c levels
Change in mean amplitude glucose excursions (MAGE | Baseline, 6 months, 12 months, 24 months
  Within and between groups difference in glucose variability measured as mean amplitude of glucose excursions (MAGE).
Change in coefficient of variation (CV) | Baseline, 6 months, 12 months, 24 months
  Within and between groups difference in glucose variability measured as coefficient of variation (CV).
Change in standard deviation (SD) of mean glucose levels | Baseline, 6 months, 12 months, 24 months
  Within and between groups difference in glucose variability measured as standard deviation (SD) of mean glucose levels
Change in glucose variability | Baseline, 6 months, 12 months, 24 months
  Within and between groups difference in time in the euglycemic range, defined as the minutes per day spent in glucose levels ranging between 70-180 mg/dL

SECONDARY OUTCOMES:
Occurrence of hypoglycemic events | Through study completion, an average of 1 year
  Number of events of mild hypoglycemia (glucose levels below 70 mg/dl), or severe hypoglycemia (below 54 mg/dl or each episode of low glucose levels requiring assistance)
Change in weight | Baseline, 12 months, 24 months
Change in lipid profile | Baseline, 12 months, 24 months
  Difference between groups in total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides
Total daily insulin doses/Kg | Baseline, 12 months, 24 months
Diabetes treatment satisfaction | Baseline, 12 months, 24 months
  In order to measure satisfaction with diabetes treatment regimens, we used the self-reported Diabetes Treatment Satisfaction Questionnaire. This instrument aims to assess levels of satisfaction in subjects using different treatment strategies. The questionnaire consists of eight questions: six questions addresses general satisfaction with a score from 0 to 6 for each question (0 = worst), that has to be computed in a total score ranging from 0 (=worst) to 36 (=best); among the remaining two questions, which has to be computed separately as two subscales, one concerns the perception of hyperglycemic events and another the perception of hypoglycemic events, both with a score from 0 (none of the time) to 6 (most of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Esposito, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Unit of Diabetes, Naples, Italy

IPD SHARING:
Plan to Share IPD: No